CLINICAL TRIAL: NCT01174199
Title: A Phase I Study of the mTOR Inhibitor Temsirolimus in Combination With the HDAC Inhibitor Vorinostat in Patients With Metastatic Prostate Cancer
Brief Title: Temsirolimus and Vorinostat in Treating Patients With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no value in finding efficacy
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPCI I 150709; NCI-2009-01537
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vorinostat; temsirolimus; Sirolimus; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral vorinostat once daily on days 1-14 and temsirolimus IV on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: temsirolimus; Other: laboratory biomarker analysis; Procedure: positron emission tomography/computed tomography

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; rapamycin analog CCI-779; Torisel
Other: laboratory biomarker analysis — Correlative study
Procedure: positron emission tomography/computed tomography — PET scan

SUMMARY:
RATIONALE: Temsirolimus and vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving temsirolimus together with vorinostat may kill more tumor cells. PURPOSE: This phase I trial is studying the side effects and best dose of temsirolimus and vorinostat in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the safety, tolerability and recommended Phase II dose of temsirolimus in combination with vorinostat in patients with metastatic, hormone refractory, chemoresistant prostate cancer. II. To obtain preliminary evidence of response in prostate cancer patients treated with temsirolimus and vorinostat. SECONDARY OBJECTIVES: I. To determine the partial and complete objective response rates in metastatic hormone-refractory, chemo-resistant prostate cancer patients with measurable disease treated with temsirolimus and vorinostat. II. To determine the progression free survival and overall survival in patients with metastatic hormone refractory, chemo-resistant prostate cancer. III. To determine the PSA response, the duration of PSA response, time to PSA progression, PSA doubling time and PSA slope in metastatic hormone refractory, chemo-resistant prostate cancer patients treated with temsirolimus and vorinostat. IV. To assess changes in expression levels of bone remodeling markers (N telopeptides and bone alkaline phosphatase) and angiogenesis-related gene and protein expression (VEGF/HIF1-alpha) in blood and circulating tumor cells, and when available, in tissue, and correlate them with cancer and treatment related outcomes. V. To assess the changes in tumor metabolism with FDG/IIC-Choline PET/CT scan. OUTLINE: Patients receive oral vorinostat once daily on days 1-14 and temsirolimus IV on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion

* Patients must have a histologically confirmed diagnosis of adenocarcinoma of the prostate that is hormone refractory and with evidence of progressive metastatic disease following docetaxel treatment by any of the following:

  * Increased serum prostate-specific antigen (PSA) levels confirmed by 3 consecutive PSA measurements (at least 2 weeks apart), the first sample to be taken at least 6 weeks after bicalutamide or megestrol acetate withdrawal AND/OR
  * Progression of bidimensionally measurable soft tissue (nodal) metastasis by CT scan or MRI within the past 4 weeks AND/OR
  * Progression of bone disease by at least two new bone lesions on bone scan confirmed by a second bone scan
* Patients should be without persisting >= grade 2 hematological/non-hematological toxicities from previous treatments that would preclude evaluation of toxic effects of study treatment.Grade 1 residual toxicity will be acceptable. Patients should be off prior therapies at least 4 weeks before starting study treatment
* Prior palliative radiation to metastatic lesion(s) is permitted, provided there is at least one measurable and/or evaluable lesion(s) that has not been radiated
* Castrate levels of serum testosterone (=< 50 ng/dL or 1.0 mmol/L) confirmed within two weeks prior to Day 1 of treatment. Testosterone levels will not be required for patients who have had bilateral orchiectomy
* ECOG performance status 0-1
* Life expectancy of greater than 6 months
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Hgb >= 9g/L
* Total bilirubin =< 1.5 x laboratory upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) <= 2.5 x laboratory ULN
* Creatinine =< 1.5 x laboratory ULN or calculated creatinine clearance >= 50 ml/min
* Serum amylase =< ULN (If > ULN, confirm pancreatic amylase < 1.1 ukat/L and serum lipase < ULN)
* PT/INR <= 1.5
* Urine protein < 1+ or if >= 1 then 24-hour urine protein should be obtained and should be < 1000 mg
* Serum cholesterol < ULN with or without treatment for hyperlipidemia; if > ULN and untreated, may be rescreened for eligibility after treatment
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of temsirolimus will be determined following review of their case by the Principal Investigator
* Patients, if sexually active, will agree to use adequate contraceptive methods (barrier contraceptive with spermicide, vasectomy, abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document
* No evidence (>= 5 years) of prior malignancies except successfully treated basal cell or squamous cell carcinoma of the skin

Exclusion

* Prior use of HDAC or mTOR inhibitors
* Patients with known brain metastases
* Any medical condition, including the presence of laboratory abnormalities, which confounds the ability to interpret data from the study or places the patient at unacceptable risk if he participates in the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or temsirolimus
* Concurrent use of other anticancer agents or treatments except LHRH antagonists
* Uncontrolled intercurrent illness including, but not limited to the following:(a)Ongoing or active infection including viral hepatitis,(b)Symptomatic congestive heart failure (New York Association Class II, III, or IV),(c) unstable angina pectoris requiring nitrate therapy,(d) prior myocardial infarction,(e)severe uncontrolled ventricular cardiac arrhythmias,(f) uncontrolled hypertension (defined as blood pressure of > 160 mmHg systolic and/or > 90 mmHg diastolic on medication),(g)electrocardiographic evidence of acute ischemia(h)Psychiatric illness/social situations that would limit compliance with study requirements
* Known positive serology for HIV and known history of HIV because of the potential for pharmacokinetic unforeseen toxicity and morbidity in an immunocompromised patient
* Any treatment modalities, including radiation and surgery, not discontinued at least 4 weeks prior to treatment in this study
* Chronic Hepatitis with advanced, decompensated hepatic disease or cirrhosis of the liver or history of chronic virus hepatitis or known viral hepatitis carrier (patient recovered from Hepatitis A will be allowed to enter the study)
* Simultaneous participation in any other study involving investigational drugs or having participated in a study less than 4 weeks prior to treatment in this study
* No investigational or commercial agents or therapies other than those described in the study may be administered with the intent to treat the patient's malignancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Frequencies of DLT and toxicity | 4 yrs
Adverse events | 4 years

SECONDARY OUTCOMES:
Median survival, median progression-free survival, and frequency of deaths | 4 years
PSA response | Every 2 cycles of treatment
Changes in expression of bone remodeling markers and angiogenesis-related gene and protein expression | Prior to each cycle
Changes in tumor metabolism as assessed by PET/CT scan | Prior to each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - The Sydney Kimmel Comprehensive Center at John Hopkins, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York